CLINICAL TRIAL: NCT01760707
Title: Exercise Capability and Training Effects in Diabetic Patients With Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9200200769; NSC92-2314-B-002-130
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus; Peripheral Neuropathy
Keywords: Diabetes mellitus; Peripheral neuropathy; Exercise; Balance performance
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Training (Experimental): aerobic exercise training
  Interventions: Behavioral: exercise training
- Control (Active Comparator)
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: exercise training
  Arms: Exercise Training
Behavioral: usual care
  Arms: Control

SUMMARY:
The purpose of the study was to investigate the effects of training on the exercise capability, balance performance, and microcirculation. Furthermore, to search the possible underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with neuropathy.

Exclusion Criteria:

* Central nerve system dysfunction, hemiparesis, motion tremor, other musculoskeletal disease that might effect the outcome measurements.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-11; Primary Completion 2003-04 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | 8 weeks
  oxygen consumption

SECONDARY OUTCOMES:
maximal oxygen pulse | 8 weeks
  maximal oxygen content in blood of each heart beat

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan